CLINICAL TRIAL: NCT06641349
Title: Effect of Maternal Multiple Micronutrient Supplementation From Preconception Through Lactation on Child Growth and Development in Rural Pakistan: A Follow-up Study
Brief Title: Effect of Maternal Supplementation From Preconception to Lactation on Child Growth and Development
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Chair, Department of Nutritional Sciences, University of Toronto
Other Study IDs: 46670
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Malnutrition; Growth &Amp; Development
Keywords: malnutrition; multiple micronutrient supplement; neurodevelopment; growth
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children born to mothers who received a multiple micronutrient supplement: From preconception to 6-months postpartum, mothers received a multiple micronutrient supplement (oral tablet at UNIMMAP composition [30 mg iron, 400 μg folic acid, 15 mg zinc, 2 mg copper, 65 μg selenium, 800 μg RE vitamin A, 1.4 mg vitamin B1, 1.4 mg vitamin B2, 18 mg niacin, 1.9 mg vitamin B6, 2.6 μg vitamin B12, 70 mg vitamin C, 5 μg vitamin D, 10 mg vitamin E and 150 μg iodine])
- Children born to mothers who received the standard of care: From preconception to 6-months postpartum, mothers received the standard of care

SUMMARY:
The goal of this observational study is to learn about the long-term effects of maternal multiple micronutrient supplementation from preconception through to lactation on child neurodevelopment and growth in a resource-limited setting where there is a high burden of malnutrition. The main questions it aims to answer are:

* Does maternal multiple micronutrient supplementation from preconception through to lactation compared to the standard of care have an effect on child neurodevelopment?
* Does maternal multiple micronutrient supplementation from preconception through to lactation compared to the standard of care have an effect on child growth?

This is a cross-sectional follow up study to a substudy of breastmilk composition and infant growth within the Matiari emPowerment and Preconception Supplementation (MaPPS) Trial, wherein mothers were randomized to receive a multiple micronutrient supplement from preconception through to lactation or the standard of care (ClinicalTrials.gov Identifier: NCT04451395).

ELIGIBILITY:
Inclusion Criteria:

* Child participated in the MaPPS Trial Breastmilk Sub-study at 3-months of age
* Child has reached their fourth birthday
* Child is available in the study catchment area (Matiari District)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residence within Matiari District, Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Full scale IQ score | At 4 years of age
  Wechsler Preschool and Primary Scale of Intelligence (WPPSI), minimum score: 40 and maximum score: 160 (higher scores mean a better outcome)

SECONDARY OUTCOMES:
Fine and gross motor skills score | At 4 years of age
  Bruininks-Oseretsky Test of Motor Proficiency, 2nd edition (BOT-2) Brief Form, minimum score: 0 and maximum score: 80 (higher scores mean a better outcome)
Height | At 4 years of age
Head circumference | At 4 years of age

OTHER OUTCOMES:
Weight | At 4 years of age
Middle upper arm circumference | At 4 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Matiari, Pakistan